CLINICAL TRIAL: NCT04467762
Title: Incidence and Severity of Neurocognitive Impairment in Pediatric Patients With Meningoencephalitis and Sepsis-associated Encephalopathy
Brief Title: Neurocognitive Impairment in Pediatric Patients With Meningoencephalitis and Sepsis-associated Encephalopathy
Acronym: NCIPED
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Johannes Ehler, MD, Principal investigator, University of Rostock
Other Study IDs: A 2020-0160
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness; Brain Injuries; Encephalopathy; Delirium; Inflammatory Disease; Central Nervous System Diseases
MeSH Terms: conditions — Critical Illness; Brain Injuries; Brain Diseases; Delirium; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and cerebrospinal fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Meningoencephalitis (ME-PED): * pediatric patients between 0 and 17 years of age
  * admission to hospital with suspected meningoencephalitis
  * confirmed meningoencephalitis within 24 hours after admission
- Sepsis-associated encephalopathy (SAE-PED): * pediatric patients between 0 and 17 years of age
  * admission to hospital with suspected sepsis
  * confirmed sepsis within 24 hours after admission or time of diagnosis
- Control group (CON-PED): * pediatric patients between 0 and 17 years of age
  * exclusion of neurocognitive impairment
  * admission to hospital for minor surgery (e.g. herniotomy, adenoidectomy, fractures treated by osteosynthesis) or for hemangioma treated by propranolol

SUMMARY:
Neurocognitive impairment is frequently observed in pediatric patients with meningoencephalitis (ME) and sepsis-associated encephalopathy (SAE) which represent two relevant central nervous system (CNS) diseases in pediatric patients. It is uncertain, if the the origin of the disease, located primarily in the CNS of patients with ME or secondarily in patients with SAE in the course of sepsis, is of importance for the severity of injury to the brain. Prospective clinical studies combining clinical and laboratory examinations including specific biomarkers of neuroaxonal injury were not performed in a comparative study. Biomarkers of neuroaxonal injury are therefore not only of great interest to detect and monitor neurocognitive impairment but also to quantify the severity of brain injury in patients with ME and SAE.

DETAILED DESCRIPTION:
This is a prospective single-center observational study evaluating the incidence and severity of the neurocognitive impairment in pediatric patients with meningoencephalitis (ME) and sepsis-associated encephalopathy (SAE). All study participants will be assessed by clinical and neurological examination as well as comprehensive laboratory tests using biomarkers of neuroaxonal injury at study day 1 (day of study inclusion), day 3 and day 5. A panel of biomarkers derived from blood and cerebrospinal fluid (CSF) samples (among others NSE, S100B and neurofilament proteins) will be measured. Clinical assessment will be performed using validated scales of severity of disease (e.g. pSOFA score) and validated delirium tests (among others pGCS, pCAM-ICU) to assess the neurocognitive performance of study participants before and three months after study inclusion (among others POPC/PCPC).

A matched group of pediatric patients without evidence for ME or sepsis/SAE will serve as a control group and will undergo the same clinical and laboratory examinations except CSF analysis.

The investigators hypothesize, that:

1. Patients with ME (primary CNS infection) indicate a higher incidence and severity of neurocognitive impairment than patients with SAE (secondary CNS affection)
2. Specific biomarkers of neuroaxonal injury in blood and CSF correlate with the clinical severity of neurocognitive impairment in patients with ME and SAE
3. Specific biomarkers of neuroaxonal injury in blood and CSF correlate with the 3-months neurocognitive outcome of patients with ME and SAE

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients between 1 day and 17 years of age
* admission to hospital with suspected meningoencephalitis or sepsis <24 hours after admission or time of diagnosis
* admission to hospital for minor surgery (herniotomy, osteosynthesis, adenoidectomy)

Exclusion Criteria:

* preexisting central nervous system diseases (stroke, hemorrhage, tumor, traumatic brain injury, brain surgery, epilepsy, hydrocephalus)
* preexisting immunosuppression
* participation in another interventional study
* no written informed consent from parents or legal representative

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients who are admitted to the study center will be screened for study eligibility according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium/neurocognitive impairment in pediatric patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | Day 90
  Assessment of neurocognitive impairment using validated tools
Change in neuroaxonal injury biomarker levels in patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | Change from baseline biomarker levels at day 5
  Measurement of biomarker levels (e.g. NSE, S100B, neurofilament proteins) derived from blood and cerebrospinal fluid samples
Neurocognitive 3-months outcome in patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | Day 90
  Assessment of the neurocognitive performance of patients using validated tests (e.g. pediatric cerebral performance category)

SECONDARY OUTCOMES:
90-day survival in patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | Day 90
  Survival after 90 days
Length of hospital stay in patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | 1 year
  Cumulative days in hospital
Length of intensive care unit stay in patients with meningoencephalitis compared to patients with sepsis-associated encephalopathy | 1 year
  Cumulative days on intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ehler, MD, Principal Investigator — University of Rostock
Locations (1):
- University Medical Center Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: No